CLINICAL TRIAL: NCT04368208
Title: Impact of Giving Birth During the Covid 19 Pandemia on Postnatal Women's Depression
Acronym: DEPRECOVID
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01065-34
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-04

CONDITIONS: Postnatal Depression
Keywords: childbirth; covid 19; satisfaction
MeSH Terms: conditions — Depression, Postpartum; COVID-19; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of postnatal depression using the the Edinburgh questionnaire between 4 and 6 weeks after delivery — The Edinburgh questionnaire is a self questionnaire validated for postnatal depression between 4 and 6 weeks postnatal
  Other Names: Assessment of satisfaction about childbirth using the WOMBLSQ4 questionnaire within the week after delivery; Retrospective assessment of prenatal anxiety within the week after the delivery; Assessment of pelvic floor disorders using the PFDI questionnaire between 4 and 6 weeks after delivery; Assessment of self rated health for the woman and the child using the WHO question about self rated health between 4 and 6 weeks after delivery

SUMMARY:
Postnatal depression is an important problematic in French population with approximatively 10 -20% of women who suffer from postnatal depression. This pathology may have strong negative impact on both women and neonate's health.

The women's satisfaction degree in front of childbirth is an important factor associated with postnatal depression since women unsatisfied of their childbirth and/or women with a complicated childbirth are more encline to suffer from postnatal depression.

It is likely that the actual context of Covid 19 pandemia and the change in obstetrical cares organization may have a negative impact on women's satisfaction about their childbirth and so a negative impact on the risk of postnatal depression.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years
* women who deliver of a singleton, term neonate in cephalic presentation

Exclusion Criteria:

* women younger than 18 years
* women who deliver of a baby in non cephalic presentation
* women with pre term Birth
* women without any internet access
* women with psychiatric disorders
* women who do not understand french language
* women who refuse to be aware of the results of the postnatal depression screening and who refuse that her doctor be ware of the results

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women who deliver of a single baby, at term and in cephalic presentation whatever is the modalities of delivery (instrumental, cesarean, spontaneous delivery) will be included after their delivery.
  Premature and non cephalic birth will be excluded because they are specific deliveries that may be assoictaed with a specific maternal anxietey. Women with psychiatric disorders are excluded since we investigated the occurrence of postnatal depression which is a psychiatric disorder.
  Women without any internet access are excluded because women will have to fill online questionnaires. Finally women will be informed, as well as their doctors, in case of postnatal depression with an advice of planning a medical consultation.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Report postnatal depression between 4 of 6 weeks during the covid 19 pandemia | 4-6 weeks postpartum
  proportion of women with an Edinburgh score higher than 12 between 4 and 6 weeks postpartum

SECONDARY OUTCOMES:
Report factors associated with postnatal depression between 4 of 6 weeks during the covid 19 pandemia | 4-6 weeks postpartum
  Existence of an association with postnatal depression and these factors: socio demographic women's characteristics, modalities of pregnancy management, satisfaction and experience about delivery, postnatal pelvic floor disorders, self rated health for the woman and the child, modalities of delivery, prenatal anxiety
Describe the experience and the satisfaction about delivery during the covid 19 pandemia | within the week after delivery
  Scale from 0 to 10 of satisfaction ; answers to the WOMBLSQ4 questionnaire about childbirth experience and satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Bertrand GACHON, Poitiers, France

IPD SHARING:
Plan to Share IPD: No